CLINICAL TRIAL: NCT02718690
Title: Importance of the Current Density: Effects of TENS About H-reflex. A Pilot Study
Brief Title: Importance of the Current Density in TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ddsm
Record Dates: First submitted 2016-03-03; First posted 2016-03-24 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2016-03

CONDITIONS: Spasticity
Keywords: H-Reflex; Current Density; TENS
MeSH Terms: conditions — Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous nerve stimulation (Experimental): Transcutaneous application of TENS current over the back for a 40 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: TENS
- Sham stimulation (Sham Comparator): Electrodes are placed over the back for a 40 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: TENS — TENS transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Transcutaneous nerve stimulation
Device: Sham stimulation — Sham transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is demonstrate the importance of density current of TENS in the effect about H-reflex in healthy volunteers.

DETAILED DESCRIPTION:
TENS have been used to treatment against pain and reflex modulation. However, the most part of evidence do not show the current density. This parameter has been demonstrated like a important factor in the effect of the current about the outcome measures.

This study show the difference between the same subjective sensation "strong but comfortable" in current density and the relation with the effect about H-reflex.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be volunteer healthy students of Physiotherapy, University of Castilla - La Mancha, older than 18 years.

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy.
* Sensitivity disturbance in lower limb.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Baseline H reflex | baseline at 0 min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
During treatment H reflex | During treatment at 33min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Post-treatment H reflex | Immediately after treatment at 40 min.
  H-reflex data are obtained by EMG signal. The EMG electrode (SignalConditioningElectrodes v2.3, Delsys Inc., USA) is fixed on triceps surae by the SENIAM protocol (www.seniam.org). The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.

SECONDARY OUTCOMES:
Change Current Density | At 1 min. treatment session, at 40 min. treatment session
  Current density (mA/cm2) is obtained by a mathematical operation. It is the result of the quotient between the current intensity by the area of the electrodes (in this case 45cm²).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos de Toledo

IPD SHARING:
Plan to Share IPD: Yes